CLINICAL TRIAL: NCT03940677
Title: Innovative Biomarkers in de Novo Parkinson's Disease
Acronym: INNOBIOPARK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: end of funding support
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Hospital, Clermont-Ferrand (Other); Grenoble Institut des Neurosciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-A02413-52
Record Dates: First submitted 2019-04-04; First posted 2019-05-07 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Parkinson's Disease; Healthy Controls Group - Age and Sex-matched
Keywords: Biomarkers; Magnetic resonance imaging (MRI); Neuropsychology; Transcranial magnetic stimulation (TMS)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson's disease patient (Other): Brain functional MRI, robotic TMS + EEG, neuropsychological evaluation, neurological examination for motor and non motor symptoms
  Interventions: Procedure: Brain MRI; Procedure: TMS-EEG; Behavioral: Behavioral and cognitive battery; Other: Clinical evaluation and clinical scales
- Healthy controls (Other): Brain functional MRI, robotic TMS + EEG, neuropsychological evaluation, neurological examination
  Interventions: Procedure: Brain MRI; Procedure: TMS-EEG; Behavioral: Behavioral and cognitive battery; Other: Clinical evaluation and clinical scales

INTERVENTIONS:
Procedure: Brain MRI — 3 Tesla brain MRI for structural and perfusion evaluation, resting state analysis and functional MRI
Procedure: TMS-EEG — Transcranial magnetic stimulation (TMS) coupled with electroencephalogram (EEG) study
Behavioral: Behavioral and cognitive battery — Emotional, attentional and behavioral assessment using predefine scales and measures
Other: Clinical evaluation and clinical scales — Neurological evaluation, ophthalmologic assessement, Montreal cognitive assessment (MoCA), movement disorder society (MDS)- UPDRS

SUMMARY:
This study aims at identifying potential new and innovative biomarkers in de novo Parkinson's disease patients. New finding will help phenotyping patients since the diagnosis of the disease and potentially also in the preclinical phase.

DETAILED DESCRIPTION:
The investigators will use 4 different approaches in parallel:

1. detailed clinical evaluation using the current available validated clinical scales and the Dopamine transporter (DAT) SPECT imaging;
2. anatomical and perfusional brain evaluation using functional MRI;
3. cortical brain mapping and transcranial magnetic stimulation assessment using a robotized approach;
4. emotional responses study using a novel paradigm. These 4 modalities will be assessed at baseline, 1 year and 2 years follow-up.

The investigators will integrate these 4 analysis using a mathematical paradigm in order to define specific phenotype of disease and disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* Asymmetric bradykinesia and/or resting tremor and rigidity since less than 2.5 years ;
* Hoehn & Yahr ≤ 2/5 ;
* Montreal cognitive assessment ≥ 26/30 ;

Exclusion Criteria:

* Treatment for Parkinson's disease (except selegiline and rasagiline)
* Severe visual/retinal pathology revealed during ophthalmological assessment
* Hyper-sensibility to gadolinium
* Renal failure
* Specific MRI contraindication
* Specific TMS contraindication

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
To compare cortical excitability differences between subjects | In a seven months period after inclusion
  The EEG data after transcranial magnetic stimulation testing will be compared between parkinsonian patients and controls
To compare brain structural differences between subjects | In a seven months period after inclusion
  All subjects will have a 3 Tesla brain MRI to collect data concerning anatomy. All data will be compared between patients and controls. Brain MRI study will consist in having the following sequences: T1 and T2, Fast Gray Matter Acquisition T1 Inversion Recovery (FGATIR)
To compare brain perfusional differences between subjects | In a seven months period after inclusion
  All subjects will have a 3 Tesla brain MRI to collect data concerning perfusion. All data will be compared between patients and controls. Brain MRI study will consist in having the following sequences: Pseudo-Continuous Arterial Spin Labeling (PCASL), T2 with gadolinium, FLAIR
To compare brain connectivity differences between subjects | In a seven months period after inclusion
  All subjects will have a 3 Tesla brain MRI to collect data concerning functional connectivity at rest. All data will be compared between patients and controls. Brain MRI study will consist in having the following sequences: Echo planar imaging (EPI) for the blood oxygen level-dependent effect
To compare emotional, attentional and behavior differences between subject | In a seven months period after inclusion
  Subjects will be asked to comment on different pictures (if the picture induces pleasure, sorrow or nothing; what would the subjects do). Attentional parameters will be recorded using the Eye tracker.
To compare emotional, attentional and behavior differences between subject with functional MRI | In a seven months period after inclusion
  During a functional MRI study, subjects will be asked to comment on different pictures (if the picture induces pleasure, sorrow or nothing; what would the subjects do). Attentional parameters will be recorded using the Eye tracker.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Moro, MD, PhD, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- CHU Grenoble Alpes, Grenoble, France